CLINICAL TRIAL: NCT02125383
Title: ParkinStim: Transcranial Direct Current Stimulation for Parkinson's Disease Phase I
Brief Title: ParkinStim: Transcranial Direct Current Stimulation for Parkinson's Disease
Acronym: ParkinStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: Rush University Medical Center (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R43NS077652-01A1 (NIH); 1R43NS077652-01A1 (NIH)
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Transcranial direct current stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Experimental): Receives 20 minutes of anodal tDCS three times while sleeping during the night.
  Interventions: Procedure: Active tDCS
- Sham tDCS (Sham Comparator): Receives 20 minutes of sham tDCS three times while sleeping during the night.
  Interventions: Procedure: Sham tDCS

INTERVENTIONS:
Procedure: Active tDCS — Anodal tDCS will be applied over motor cortex for 20 minutes, three times during the night while the subject sleeps, each separated by 1 hour
  Arms: Active tDCS
Procedure: Sham tDCS — Sham tDCS will be applied over motor cortex for 20 minutes, three times during the night while the subject sleeps, each separated by 1 hour
  Arms: Sham tDCS

SUMMARY:
The purpose of this study is to evaluate the effects of transcranial direct current stimulation (tDCS) on patients with Parkinson's disease during sleep.

DETAILED DESCRIPTION:
The clinical study will follow a counterbalanced crossover design during which subjects will undergo two separate pairs of two-consecutive-overnight sleep studies and receive anodal tDCS (active or sham) to M1. The first sleep study in each pair will acclimate subjects to the sleep laboratory and minimize "first night" effects, thus no tDCS will be applied. The second sleep study in each pair will include active or sham tDCS, presented in a pseudorandom order such that approximately half of the subjects receive active tDCS first while the other half receives sham first. The two pairs of sleep studies will be separated by one to three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's disease (PD) according to the UK PD brain bank criteria
* Hoehn and Yahr stage II-III when off anti-parkinsonian medication
* Able to provide informed consent
* Currently taking levodopa (300-800 mg per day)
* On stable regimen of anti-parkinsonian medication for at least one month before study entry and able to continue on a stable regimen for the duration of the study
* Presence of early morning akinesia
* Naïve to tDCS.

Exclusion Criteria:

* Children will be excluded from this study due to the fact that they are unlikely to have PD
* Significant medical or psychiatric illness, significant neurological disease other than PD, metal objects and/or deep brain stimulators in the head that might pose a hazard during tDCS
* Dementia, as evidenced by a score less than 26 on the Montreal Cognitive Assessment
* Significant depression (Geriatric Depression Scale score < 20)
* Presence of hallucinations
* Having undergone any surgical procedure for treatment of PD including deep brain stimulation (DBS), pallidotomy, thalamotomy, or other brain surgeries
* A history of seizures
* A known history of severe sleep apnea or sleep onset insomnia
* Skin diseases that could potentially cause irritations under electrodes

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
PD motor scores measured by Kinesia HomeView | Average change from two days before tDCS sleep study to two days after tDCS sleep study
  PD motor symptoms will be assessed for two days before (baseline) and two days after each tDCS sleep study using Kinesia HomeView. Changes for active tDCS will be compared to changes for sham tDCS.

SECONDARY OUTCOMES:
Sleepiness | Average change from two days before tDCS sleep study to two days after tDCS sleep study
  Epworth Sleepiness Scale
tDCS sensations | Day after tDCS sleep studies
  Each subject will complete a questionnaire regarding sensations they felt during the night the day after each tDCS sleep study.
Motor scores measured by the Unified Parkinson's Disease Rating Scale | Average change from day before tDCS sleep study to day after tDCS sleep study
Overnight Polysomnography | During each sleep study
  Polysomnography parameters will be compared during the active and sham tDCS sleep studies.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin A Heldman, Ph.D., Principal Investigator — Great Lakes NeuroTechnologies
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States